CLINICAL TRIAL: NCT02082379
Title: In-Vivo Evaluation of Nebulized Aerosols Delivered Via Nasal Route
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 202438
Record Dates: First submitted 2014-02-11; First posted 2014-03-10 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Interface Acceptance During Delivery of Aerosol Medicine to an Infant or Child
Keywords: Interface, aerosol, child, acceptance

ARMS (2):
- Term newborns 1-6 week old (Active Comparator): A Hudson nebulizer will be loaded with 3 mls of normal saline and operated at 7 L/min of wall air for 3 minutes with each scenario with a 5-minute interval between interfaces. The interfaces that will be used are: tight mask, the angled PediNeb, the B&B adapter, mask placed at 2 cm from the face, the PediNeb T-piece, and a capped corrugated tubing placed 2 cm away from the face.
  Interventions: Behavioral: inhaled normal saline using different interfaces.
- Infants 6-8 month old (Active Comparator): A Hudson nebulizer will be loaded with 3 mls of normal saline and operated at 7 L/min of wall air for 3 minutes with each scenario with a 5-minute interval between interfaces. The interfaces that will be used are: tight mask, the angled PediNeb, the B&B adapter, mask placed at 2 cm from the face, the PediNeb T-piece, and a capped corrugated tubing placed 2 cm away from the face.
  Interventions: Behavioral: inhaled normal saline using different interfaces.

INTERVENTIONS:
Behavioral: inhaled normal saline using different interfaces. — A Hudson nebulizer will be loaded with 3 mls of normal saline and operated at 7 L/min of wall air for 3 minutes with each scenario with a 5-minute interval between interfaces. The infants will be videotape while they receive inhaled aerosol, and sound will be captured. The camera will be positioned so the face of the parent holding the child will not be visible.

SUMMARY:
We hypothesize that infant and children will show different levels of acceptance of different interfaces while they receive inhaled therapy.

We also hypothesize that children will exhibit different amounts of time with the aerosol well aligned with the nostrils during transnasal aerosol delivery.

DETAILED DESCRIPTION:
Aerosol medicine is widely used in treating pulmonary diseases in children. Delivering drugs via aerosol faces several challenges; some are related to the drug and the delivery methods and others to the patient behavior. The latter are crucial and can significantly affect the lung deposition of the drug. Infants are known to be obligate nose breathers making the transnasal route the natural approach for drug delivery in this age group. Different interfaces are already available in the market and are specifically designed to be used in children to improve the child acceptability of the interface and by the result to improve drug deposition. Due to limitations in the use of radiolabeled aerosols and pharmacokinetics/pharmacodynamics studies in infants and children, in-vitro models were developed. These models still lack biological variability which leads to overestimating lung deposition. So, real life correction factors are needed to improve current in-vitro modeling. Previous unpublished data from our laboratory showed that alignment of the aerosol stream with the nostrils is very important for pulmonary deposition.

Our objectives are to provide real life data of acceptance of different interfaces by infants and children and to provide a real life correction factor to improve current in-vitro modeling.

ELIGIBILITY:
Inclusion Criteria:

* Born at term
* Healthy
* Pacifier user
* Newborn 1-6 week old
* Infants 6-8 month old

Exclusion Criteria:

* Chronic respiratory disease
* Cardiac disease
* Prematurity
* Neurological disease
* Allergy to Normal Saline
* Allergy to any components of the interfaces

Ages: 1 Week to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Acceptance of different interfaces while they receive inhaled therapy | within the 3 minutes of nebulization for 3 consecutive times with 5 minutes rest in between the each nebulization
  The recordings will be analyzed by the 2 investigators for acceptance of the patient of the interface (likert scale 1 to 5: 5= Complete acceptance, 4= Accepting most of the time, 3= Accepting/rejecting half of the time, 2= Rejecting most of the time, 1= Complete rejection). The data will be expressed as average of value assigned by each of the 2 researchers. Analysis of variance for repeated measures followed by Tukey test will be used to compare the 2 endpoints. A p value < 0.05 will be considered statistically significant

SECONDARY OUTCOMES:
Amounts of time with the aerosol well aligned with the nostrils during transnasal aerosol delivery | during the 3 minutes of nebulization
  The recordings will be analyzed by the 2 investigators for percentage of time spent with aerosol aligned with the patient nostrils when using different interfaces

CONTACTS AND LOCATIONS:
Overall Officials: Katia El Taoum, MD, Principal Investigator — UAMS; Ariel Berlinski, MD, Principal Investigator — UAMS/ACHRI
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States